CLINICAL TRIAL: NCT05855083
Title: A Phase 2 Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Narsoplimab in Pediatric Patients (28 Days to ≤ 18 Years of Age.) With High-Risk Hematopoietic Stem Cell Transplant Thrombotic Microangiopathy
Brief Title: Efficacy and Safety Study of Narsoplimab in Pediatric Patients With High-Risk Hematopoietic Stem Cell Transplant TMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS721-HCT-002
Expanded Access: NCT04247906 (Available)
Record Dates: First submitted 2023-04-06; First posted 2023-05-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Thrombotic Microangiopathies; Hematopoietic Stem Cell Transplantation
Keywords: TMA; HSCT; Pediatric; BMT; OMS721; Narsoplimab
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — narsoplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Narsoplimab single arm-treatment (Experimental): Narsoplimab 4 mg/kg
  Interventions: Drug: Biological: narsoplimab

INTERVENTIONS:
Drug: Biological: narsoplimab — Treatment with narsoplimab 4 mg/kg will be administered
  Other Names: Narsoplimab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of narsoplimab in pediatric patients with thrombotic microangiopathies (TMA) following hematopoietic stem cell transplant (HSCT).

DETAILED DESCRIPTION:
This is a Phase 2, uncontrolled, single-dosing regimen study in pediatric patients from 28 days to less than 18 years of age with high risk HSCT-TMA. At least 4 patients will be required from each of 3 age cohorts:

28 days to <2 years of age, 2 years to <12 years of age, and 12 years to <18 years of age.

Treatment will be for 8 weeks and patients will be followed for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 28 days and less than 18 years prior to informed consent (Visit 0).
2. Have informed consent from at least one parent or legal guardian as required by local law and regulation. Patient informed consent will be required if the patient has reached the local legal age of majority.
3. Assent from patients as required by local law and regulation.
4. Have received an allogeneic hematopoietic stem cell transplant for the treatment of benign or malignant disease.
5. Have a diagnosis of HSCT-TMA defined as meeting both of the following criteria:

   * Platelet count < 50,000/mL or a decrease in platelet count > 50% from the highest value obtained following transplant.
   * Evidence of microangiopathic hemolysis (presence of schistocytes, serum lactate dehydrogenase [LDH] > upper limit of normal ([ULN], or haptoglobin < lower limit of normal [LLN])
6. Have at least one of the following HSCT-TMA high-risk criteria:

   * HSCT-TMA persistence > 2 weeks following modification of calcineurin inhibitors or sirolimus OR
   * Have evidence of high-risk HSCT-TMA defined as at least one of the following:

     * Spot protein/creatinine ratio > 2 mg/mg
     * Serum creatinine > 1.5 x the creatinine level prior to TMA development
     * Biopsy-proven gastrointestinal TMA
     * TMA-related neurological abnormality
     * Pericardial or pleural effusion without alternative explanation
     * Pulmonary hypertension without alternative explanation
     * Have Grade III or Grade IV graft-versus-host disease (GVHD) or, in the opinion of the Investigator, risk for development of Grade III or Grade IV GVHD if immunosuppression were to be modified
     * Have elevated serum C5b-9 (> 244 ng/mL)
7. If sexually active and of childbearing potential (for female pediatric patients, defined as starting at onset of menses), must agree to practice a highly effective method of birth control throughout study drug treatment and for at least 12 weeks after the last dose of study drug, such method of birth control defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence (abstinence is acceptable when it is in line with the patient's preferred and usual lifestyle and is defined as complete abstinence of sexual intercourse, not periodic abstinence or withdrawal), or vasectomized partner.
8. Male patients must be willing to avoid fathering children for at least 12 weeks following the last dose of study medication.

Exclusion Criteria:

1. All treatments for HSCT-TMA are allowed except eculizumab, ravulizumab, and defibrotide within 3 months prior to informed consent, unless failure of therapy can be documented.

   a. Patients may not be on eculizumab, ravulizumab, or defibrotide for any indication at screening.
2. Have Shiga toxin-producing Escherichia coli haemolytic uraemic syndrome (STEC-HUS). Test results obtained within 28 days prior to informed consent may be used.
3. Have ADAMTS13 activity < 10%. Test results obtained within 28 days prior to informed consent may be used.
4. Have a severe, uncontrolled systemic bacterial or fungal infection requiring antimicrobial therapy, or a severe uncontrolled viral infection (as determined by the investigator); prophylactic antimicrobial therapy administered as standard of care is allowed.
5. Have malignant hypertension (blood pressure [BP] > 99th percentile plus 5 mmHg with bilateral hemorrhages or "cotton-wool" exudates on fundoscopic examination).
6. Due to conditions other than HSCT-TMA, have a poor prognosis with a life expectancy of less than 3 months in the opinion of the Investigator.
7. If pregnant or lactating.
8. Have received treatment with an investigational drug or device within 4 weeks of entering study.
9. Have abnormal liver function tests defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times ULN within 28 days prior to informed consent.
10. Have a positive test by antigen or polymerase chain reaction (PCR) for human immunodeficiency virus (HIV), if negative within 28 days prior to informed consent, the test does not need to be repeated.
11. Patient or one or more of the patient's parents or legal guardians are is an employee or an immediate family member of Omeros, the Clinical Research Organization (CRO), an Investigator, or a study staff member.
12. Have a known hypersensitivity to any constituent of the product.
13. Presence of any condition that the Investigator believes would put the patient at risk.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
100-day survival rate following high-risk HSCT-TMA diagnosis. | 100 days
  Percentage of patients alive at 100 days following the diagnosis of high-risk HSCT-TMA

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events assessed by CTCAE v5.0 | 52 weeks
  Number and percentage of patients with treatment-emergent adverse events will be summarized by MedDRA system organ class and preferred term
Percentage of patients meeting protocol definition of clinical response | 52 weeks
  A responder is defined as a patient with HSCT-TMA who demonstrates improvement in laboratory TMA markers (platelet count and LDH) and clinical benefit (either improvement in organ function or reduction in transfusion burden)
52 week survival rate following high-risk HSCT-TMA diagnosis | 52 weeks
  Percentage of patients alive at 52 weeks following the diagnosis of high-risk HSCT-TMA
Overall survival following the diagnosis of high-risk HSCT-TMA | 52 weeks
  Median overall survival (days) following the diagnosis of high-risk HSCT-TMA by Kaplan-Meier estimate
Pharmacokinetics (PK) of multiple-dose administration of OMS721 | 52 weeks
  PK parameters including maximum concentration and minimum (trough) concentration
Presence of anti-drug antibody (ADA) | 52 weeks
  Number and percentage of patient with at least one ADA positive sample

CONTACTS AND LOCATIONS:
Locations (16):
- United States (8):
  - Omeros Investigational Site, San Diego, California
  - Omeros Investigational Site, Gainesville, Florida
  - Omeros Investigational Site, Boston, Massachusetts
  - Omeros Investigational Site, St Louis, Missouri
  - Omeros Investigational Site, New York, New York
  - Omeros Investigational Site, Valhalla, New York
  - Omeros Investigational Site, Houston, Texas
  - Omeros Investigational Site, Seattle, Washington
- Germany (2):
  - Omeros Investigational Site, Halle
  - Omeros Investigational Site, Hanover
- Israel (4):
  - Omeros Investigational Site, Haifa
  - Omeros Investigational Site, Jerusalem
  - Omeros Investigational Site, Ramat Gan
  - Omeros Investigational Site, Tel Aviv
- Omeros Investigational Site, Utrecht, Netherlands
- Omeros Investigational Site, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No